CLINICAL TRIAL: NCT01220024
Title: A Phase II, Randomized, Single Dose, Double-blind, Placebo Controlled Study to Investigate the Efficacy and Safety Profile of the CollaRx® Bupivacaine Implant (200 mg Bupivacaine Hydrochloride) in Men After Open Laparotomy Herniorrhaphy
Brief Title: Safety and Efficacy of CollaRx® Bupivacaine Implant in Men After Open Laparotomy Herniorrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INN-CB-010
Record Dates: First submitted 2010-09-23; First posted 2010-10-13 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Herniorrhaphy; Postoperative Pain; Inguinal Hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Bupivacaine; Collagen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2, 5x5cm bupivacaine collagen sponges (Experimental): collagen sponges
  Interventions: Drug: Bupivacaine Collagen Sponge
- 2, Placebo collagen sponges (Placebo Comparator): Placebo collagen sponges
  Interventions: Drug: Placebo collagen Sponge

INTERVENTIONS:
Drug: Bupivacaine Collagen Sponge — Drug: Bupivacaine Collagen Sponge
  Other Names: Bupivacaine Implant
  Arms: 2, 5x5cm bupivacaine collagen sponges
Drug: Placebo collagen Sponge — Drug: Placebo Collagen Sponge
  Other Names: Collagen Implant
  Arms: 2, Placebo collagen sponges

SUMMARY:
This study will assess pain intensity for the first 72 hrs after after aggravated movement (cough)following open laparotomy inguinal herniorrhaphy in patient who receive either the CollaRx Bupivacaine implant or a plain collagen sponge.

DETAILED DESCRIPTION:
Inguinal herniorrhaphy is a common surgery; and common surgical methods used include laparoscopic and open placement of synthetic mesh. The use of synthetic mesh can greatly reduce the risk of hernia recurrence regardless of the method used for its placement. Managing postoperative pain and preventing morbidity after open mesh herniorrhaphy remain considerable medical challenges.

Bupivacaine is a local anesthetic (pain medicine) that has an established safety profile. Collagen is a protein that is found in all mammals. The CollaRx Bupivacaine implant is a thin flat sponge made out of collagen that comes from cow tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the site but very little is absorbed into the blood stream. The high levels of bupivacaine at the surgical site may result in less pain for several days after surgery.

This study will assess pain intensity after surgery in patients who receive either the CollaRx Bupivacaine implant or a plain collagen sponge.

ELIGIBILITY:
Inclusion Criteria:

* Man ≥ 18 years
* Body mass index (BMI) ≥ 19 and ≤ 40 kg/m2.
* Has a planned unilateral inguinal herniorrhaphy (open laparotomy, tension free technique) to be performed according to standard surgical technique under general anesthesia.

Exclusion Criteria:

* Has a known hypersensitivity to amide local anesthetics, opioids, or bovine products.
* Scheduled for bilateral inguinal herniorrhaphy.
* Undergone a prior herniorrhaphy on the side scheduled for repair.
* Undergone major surgery within 3 mos of the scheduled herniorrhaphy.
* Has cardiac arrhythmias or atrioventricular (AV) conduction disorders.
* Concomitantly uses antiarrhythmics (eg, amiodarone, lidocaine), propranolol, or strong/moderate cytochrome P450 (CYP) 3A4 inhibitors or inducers (eg, macrolide antibiotics and grapefruit juice).
* Used long acting analgesics within 24 hours of surgery. Short acting analgesics such as acetaminophen may be used on the day of surgery but are subject to preoperative restrictions for oral intake.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2011-05-18 (Actual); Study Completion 2011-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Bellaire, Texas, United States

REFERENCES:
- [Result] Cusack SL, Jaros M, Kuss M, Minkowitz HS, Winkle P, Hemsen L. Clinical evaluation of XaraColl((R)), a bupivacaine-collagen implant, for postoperative analgesia in two multicenter, randomized, double-blind, placebo-controlled pilot studies. J Pain Res. 2012;5:217-25. doi: 10.2147/JPR.S33453. Epub 2012 Jun 27. PMID 22792007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical investigative sites
Groups:
- 2, 5x5cm Bupivacaine Collagen Sponges: Bupivacaine Collagen Sponge: Drug: Bupivacaine Collagen Sponge - Two 5 × 5-cm bupivacaine sponges each containing 75 mg of Type I collagen and 100 mg bupivacaine hydrochloride,
- 2, Placebo Collagen Sponges: Placebo collagen Sponge: Drug: Placebo Collagen Sponge - Two 5 × 5-cm placebo sponges each containing 75 mg of Type I collagen.
Period: Overall Study
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.3) | 41.7 (14.9) | 44.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Defined as Area Under the Curve (AUC) of 100-mm VAS PI Scores.
Description: The primary efficacy variable was SPI defined as area under the curve (AUC) of 100-mm VAS pain intensity scores after aggravated movement (cough) from 1 to 72 hours after surgery. Minimum score is "0". Maximum score is 7200. This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule. A lower score means a better outcome or less pain reported.
Time Frame: 1, 2, 4, 6, 8, 10, 12, 24, 48, and 72 hours.
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: score on a scale*hour
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Number analyzed (Participants) | 25 | 24
score on a scale*hour | 2810.4 (1693.43) | 3484.5 (1806.68)

2. Secondary Outcome: Sum of Pain Intensity (SPI) After Aggravated Movement (Cough)
Description: Measured on a Visual Analog Pain Scale (VAS) with the lowest possible value of 0 and highest 100 (0 - 100) at each time point. A lower score is better which means the patient experience lower pain. The score is calculated using the number of hours * the VAS score. This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule. For each measure outcome - the minimum score is "0" and the maximum score is 100* the number of hours in that period.
Time Frame: 1, 2, 4, 6, 8, 10, 12, 24, 48, and 72 hours.
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale*hour
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Number analyzed (Participants) | 25 | 24
score on a scale*hour
  1 to 24 hours | 996.3 (503.65) | 1270.4 (566.52)
  25 to 48 hours | 1021.8 (604.71) | 1186.7 (647.40)
  1 to 48 hours | 2018.2 (1092.85) | 2457.2 (1155.63)
  49 to 72 hours | 792.2 (633.88) | 1027.4 (713.60)

3. Secondary Outcome: Sum of Pain Intensity (SPI) Using a Visual Analog Scale (VAS) When at Rest
Description: as for outcome 2
Time Frame: 1, 2, 4, 6, 8, 10, 12, 24, 48, and 72 hours.
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale*hour
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Number analyzed (Participants) | 25 | 24
score on a scale*hour
  1 to 24 hours | 741.6 (452.29) | 856.6 (486.95)
  25 to 48 hours | 754.7 (538.41) | 677.2 (455.96)
  1 to 48 hours | 1496.4 (978.74) | 1533.8 (875.52)
  49 to 72 hours | 567.0 (565.64) | 501.3 (451.92)
  1 to 72 hours | 2063.4 (1511.89) | 2035.0 (1271.12)

4. Secondary Outcome: Pain Intensity Visual Analog Pain Scale Scores Over Time After Aggravated Movement (Cough)
Description: Measured on a Visual Analog Pain Scale (VAS) with the lowest possible value of 0 and highest 100 (0 - 100). Patients were asked during multiple time points to provide a score on this VAS scale. The lower the sore the better the outcome. Higher score is a worse outcome
Time Frame: 1,2,4,6,8,10,12,24,48 and 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Number analyzed (Participants) | 25 | 24
units on a scale
  Hour 1 | 31.4 (28.59) | 73.4 (22.61)
  Hour 2 | 32.6 (24.88) | 60.6 (22.81)
  Hour 4 | 31.2 (26.10) | 57.0 (24.79)
  Hour 6 | 33.2 (24.95) | 58.8 (26.05)
  Hour 8 | 47.0 (24.83) | 54.3 (27.49)
  Hour 10 | 43.4 (25.54) | 52.0 (30.41)
  Hour 12 | 46.7 (28.18) | 28.18 (29.72)
  Hour 24 | 49.2 (26.37) | 51.5 (26.65)
  Hour 48 | 36.0 (27.31) | 47.2 (29.78)
  Hour 72 | 29.8 (27.00) | 38.3 (30.16)

5. Secondary Outcome: Pain Intensity VAS Scores Over Time at Rest
Description: Measured on a Visual Analog Pain Scale (VAS) with the lowest possible value of 0 and highest 100 (0 - 100). Patients were asked during multiple time points to provide a score on this VAS scale. Lower score is better. Higher score means more pain. Time points are summarized independently
Time Frame: 1,2,4,6,8,10,12,24,48 and 72 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Number analyzed (Participants) | 24 | 24
score on a scale
  Hour 1 | 31.6 (29.20) | 73.4 (22.61)
  Hour 2 | 33.2 (25.20) | 60.6 (22.81)
  Hour 4 | 31.6 (24.60) | 57.0 (24.79)
  Hour 6 | 33.5 (25.45) | 58.8 (26.05)
  Hour 8 | 47.3 (25.33) | 54.3 (27.49)
  Hour 10 | 44.0 (25.93) | 52.0 (30.41)
  Hour 12 | 47.6 (28.47) | 55.2 (29.72)
  Hour 24 | 49.3 (26.92) | 51.5 (26.65)
  Hour 48 | 36.3 (27.85) | 47.2 (29.78)
  Hour 72 | 30.7 (27.23) | 38.3 (30.16)

6. Secondary Outcome: Mean Sum of Pain Intensity (SPI) Categorical Scores After Aggravated Movement
Description: Measured on a Visual Analog Pain Scale (VAS) with the lowest possible value of 0 and highest 100 (0 - 100) for each timepoint. (timepoints 1,2,4,6,8,10,12,24,48 and 72 hours ) Patients were asked during multiple time points to provide a score on this VAS scale. For 1 to 24 hours the highest score possible would be 800. For 1 to 48 hours the highest score possible would be 900. For 1 to 72 hours the highest score possible would be 1000. A mean Lower score is better. A mean Higher score is a worse outcome.
Time Frame: 1,2,4,6,8,10,12,24,48 and 72 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
Number analyzed (Participants) | 25 | 24
score on a scale
  1 to 24 hours | 40.6 (13.64) | 45.6 (13.84)
  1 to 48 hours | 83.3 (29.63) | 90.2 (27.86)
  1 to 72 hours | 118.9 (44.80) | 128.8 (46.12)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 2, 5x5cm Bupivacaine Collagen Sponges | 2, Placebo Collagen Sponges
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 15/25 | 17/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2, 5x5cm Bupivacaine Collagen Sponges (N=25) | 2, Placebo Collagen Sponges (N=25)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chills (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Incision site infection (Infections and infestations) | 2 (2) | 0 (0) — both were mild
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Scrotal swelling (Reproductive system and breast disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other